CLINICAL TRIAL: NCT01844648
Title: A Randomized, Double-blind, Placebo-controlled, Crossover Study of the Safety and Efficacy of Tropicamide 1 mg Intra-oral Slow Dissolving Muco-adhesive Thin Films to Reduce Hypersalivation in PD Patients Manifesting Sialorrhea Complaints
Brief Title: Study of the Safety and Efficacy of Tropicamide Thin Films to Reduce Hypersalivation in Parkinson's Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroHealing Pharmaceuticals Inc. (Industry)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NH004-3; 2011-004212-36 (EudraCT Number)
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2014-04

CONDITIONS: Sialorrhea (Excessive Drooling)
Keywords: Parkinson's disease; Sialorrhea; Tropicamide; Non-motor symptoms; Thin strip delivery
MeSH Terms: conditions — Sialorrhea; Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NH004 tropicamide (Experimental): tropicamide 1 mg thin film, twice daily for 7 days
  Interventions: Drug: NH004 tropicamide
- NH004 placebo (Placebo Comparator): placebo thin film, twice daily for 7 days
  Interventions: Drug: NH004 Placebo

INTERVENTIONS:
Drug: NH004 tropicamide — Intra-oral slow dissolving muco-adhesive thin film containing 1 mg tropicamide
  Arms: NH004 tropicamide
Drug: NH004 Placebo — Intra-oral slow dissolving muco-adhesive thin film
  Arms: NH004 placebo

SUMMARY:
To study the safety and efficacy of tropicamide 1 mg intra-oral slow dissolving muco-adhesive thin films compared to placebo to reduce hypersalivation in PD patients manifesting sialorrhea complaints.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomized, crossover, multicentre study comparing intra-oral slow dissolving muco-adhesive thin films containing tropicamide 1 mg or Placebo. Patients will receive each treatment twice daily (1 h after breakfast and 1 h after lunch) for 1-week.

Patients will be evaluated for eligibility during the 14-day screening period. Those patients meeting all entry criteria at baseline will be randomized (1:1) to receive first tropicamide followed by placebo films or vice versa. Patients will return for regularly scheduled visits at Weeks 1 and 3 or at early discontinuation.

ELIGIBILITY:
Inclusion criteria:

* Patients with idiopathic Parkinson's disease, according to the UK Brain Bank criteria.
* Patients complaining of drooling, with a score of at least 6 points in the SCS-PD scale.
* Patients above 30 years old.
* Patients with Hoehn & Yahr score between I-IV.
* Male or non-pregnant female. Females of child-bearing potential will be required to have undergone a pregnancy test with negative results prior to entry to the study and agree to use contraceptive measures for the duration of the study.
* Patients must have used the same antiparkinsonian medications and at the same dose for the last month. No changes in the medication for PD are expected during the study.

Exclusion criteria:

* Pregnant women.
* Patients with a secondary parkinsonian syndrome, parkinsonism-plus syndromes, heredodegenerative disorders or benign parkinsonism.
* Patients with a diagnosis of major depression or psychosis according to the DSM-IV.
* Patients with MMSE score equal to or lower than 24.
* Patients with a current diagnosis of substance abuse (DSM-IV) or history of alcohol or drug abuse in the past 3 months.
* Patients with hallucinations.
* Patients with a current clinically significant gastrointestinal, renal, hepatic, endocrine, pulmonary or cardiovascular disease, including hypertension that is not well-controlled, asthma, chronic obstructive pulmonary disease (COPD) and Type I diabetes.
* Patients with a second- or third-degree atrioventricular block or sick sinus syndrome, uncontrolled atrial fibrillation, severe or unstable angina, congestive heart failure, myocardial infarction within 3 months of the screening visit, or significant ECG abnormality, including QTc ≥ 450 msec (males) or ≥ 470 msec (females), where QTc is based on Bazett's correction method.
* Patient with a neoplastic disorder, which is either currently active or has been in remission for less than one year.
* Patients with a history or a current diagnosis of HIV, or tests positive for Hepatitis B or C antibodies, or Hepatitis B surface antigen
* Patients who have participated in a previous clinical trial within 30 days of entry into the study (screening visit) or have received treatment with any investigational compound within 30 days.
* Patients with hypersensitivity to atropine or other anticholinergic drugs.
* Patients who have experienced adverse effects as a result of taking anticholinergic drugs.
* Patients who are receiving any anticholinergic drug or an anticholinesterase agent.
* Patients who started or changed the dose of any of the following medications in the previous week: tricyclic antidepressants, monoamine oxidase-A inhibitors, antipsychotics, benzodiazepines, opioids, antihistamines, carbamazepine, NSAIDs.
* Patients with significant dental/oral pathology.
* Patient with any abnormality that the investigator deems to be clinically relevant, either on medical history, physical examination, ECG or in a diagnostic laboratory test.
* Patients with closed-angle Glaucoma or those at high risk of suffering it after treatment with anticholinergic agents.
* Patients with Prostatic Adenoma.
* In the judgment of the Clinical Investigator, the patient is likely to be non-compliant or uncooperative during the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
modified Teachers Drooling Scale (% responding) | one week
  The primary endpoint for this trial is the difference in responder rate between tropicamide and placebo. Responders will be defined as subjects whose mean sialorrhea score improved by at least 30% as compared to baseline in the 9-point modified Teachers Drooling Scale (mTDS).

SECONDARY OUTCOMES:
modified Teachers Drooling Scale (mean) | one week
  Difference in the mean sialorrhea scores between placebo and tropicamide in the 9-point modified Teachers Drooling Scale (mTDS).
Sialorrhea Clinical Scale for Parkinson's Disease (mean) | one week
  - Difference in the mean sialorrhea scores between placebo and tropicamide in the Sialorrhea Clinical Scale for Parkinson's Disease (SCS-PD).
UPDRS Part II sialorrhea item (mean) | one week
  Difference in the mean sialorrhea scores between placebo and tropicamide in the UPDRS Part II sialorrhea item (#6).
Visual Analg Scale | one week
  Saliva buccal content as measured by a Visual Analog Scale (VAS) score, evaluated before and during 3 hours after treatments administration.

CONTACTS AND LOCATIONS:
Overall Officials: Elkan R Gamzu, PhD, Study Director — NeuroHealing Pharmaceuticals Inc.
Locations (3):
- France (3):
  - Hôpital de la Salpêtrière, Paris, Cedrex 13
  - Hôpital Paul de Viguier, Toulouse, Cedrex 9
  - Hôpital Haut Lévêque, Bordeaux, Pessac